CLINICAL TRIAL: NCT02427009
Title: Effectiveness of Maintaining a Prone Position After Use of an Epidural Blood Patch for the Treatment of Post-dural Puncture Headache
Brief Title: Maintaining a Prone Position After Use of an Epidural Blood Patch for the Treatment of Post-dural Puncture Headache
Acronym: UpSideDown
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no inclusion
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LOCAL/2015/GA-01; 2014-A01921-46 (Other: RCB number)
Record Dates: First submitted 2015-04-20; First posted 2015-04-27 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Post-Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Prone Position; Blood Patch, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The study population (Experimental): The study population consists of adult women requiring an epidural blood patch for the treatment of post-dural puncture headache following vaginal delivery. Women who delivered by cesarean section are not included due to the discomfort of the prone position while there is an abdominal scar.
  Intervention: Prone position for 1 hour after blood patch
  Interventions: Other: Prone position for 1 hour after blood patch; Procedure: Blood patch

INTERVENTIONS:
Other: Prone position for 1 hour after blood patch — After performing a blood patch, the patient will be placed in a prone position for 1 hour. This applies to all blood patches required during her hospitalization.
Procedure: Blood patch — And indicated in inclusion criteria, patients in this protocol will have at least 1 blood patch. The amount of blood to be injected into the peridural space is fixed at 20 ml, but can be less in case of pain.

SUMMARY:
The main objective of this study is to assess the rate of recurrence of headache following a first blood patch where patients will be positioned in the prone position for an hour after each blood patch needed during this study.

DETAILED DESCRIPTION:
The secondary objectives of this study are to:

A. To evaluate the number of blood patches needed for each patient during her hospital stay B. Assessing the intensity of all headaches every 24H C. Evaluate the complications occurring during the hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* The patient was informed about the implementation of the study, its objectives, constraints and patient rights
* The patient has signed the informed consent
* The patient must be affiliated or beneficiary of a health insurance plan
* The patient is available for follow up concerning her hospital stay
* The patient has a post-dural puncture headache after a vaginal delivery. The diagnosis of post-puncture headache is retained on the basis of a frankly postural character for the headache, triggered or exacerbated by orthostatic position and relieved by recumbency.
* The patient has an indication for a blood patch

Exclusion Criteria:

* The patient is participating in another interventional study, with the exception of the following studies: Papillo PMA (2013-A00538-37); DG-Postpartum (2013-A00277-38); ElastoMAP (2013-A01148-37); ElastoDéclench (2014-A00828-39); LXRs(2009-A00968-49); OASIS II (2013-A00773-42); GrossPath (2014-A01120-47).
* The patient is in an exclusion period determined by a previous study
* The patient is under guardianship, curatorship or under judicial protection
* The patient refuses to sign the consent
* It is not possible correctly inform the patient
* The patient is pregnant
* The patient has a contra-indication (or an incompatible combination therapy) for a necessary treatment in this study
* The patient was delivered by cesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04-21 (Actual); Study Completion 2016-04-23 (Actual)

PRIMARY OUTCOMES:
Headache recurrence: yes/no | 24 hours after first blood patch
  Headache recurrence defined by: presence of headaches that confine the mother to bed or affect her ability to take care of her baby
Headache recurrence: yes/no | 48 hours after first blood patch
  Headache recurrence defined by: presence of headaches that confine the mother to bed or affect her ability to take care of her baby
Headache recurrence: yes/no | 72 hours after first blood patch
  Headache recurrence defined by: presence of headaches that confine the mother to bed or affect her ability to take care of her baby

SECONDARY OUTCOMES:
The number of blood patches required for each patient | Hospital discharge (expected average of 7 days)
Visual analog scale for pain | Baseline (day 0)
  Scale from 0.0 to 10.0.
Visual analog scale for pain | 24 hours after blood patch
  Scale from 0.0 to 10.0.
Visual analog scale for pain | 48 hours after blood patch
  Scale from 0.0 to 10.0.
Visual analog scale for pain | 72 hours after blood patch
  Scale from 0.0 to 10.0.
Presence/absence of complications | During hospital stay (expected average of 7 days)
  Presence / absence of the following complications: nerve paresthesia; nerve damage; accidental dural puncture; subcutaneous hematoma at the puncture site; meningitis; epidural abscess; localized infection at the puncture site; encephalopathy; cerebral venous thrombosis; subdural hematoma
In case of recurrence of headache following the 1st blood patch, the presence / absence of the following accompanying symptoms: nausea; vomiting; dizziness; tinnitus; diplopia; photophobia; low back pain. | During hospital stay (expected average of 7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Aya, MD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France